CLINICAL TRIAL: NCT06135597
Title: Role of Cellular Immune Regulation in Acute Exacerbation and Chronic Aspergillus Infection After COVID-19 Infection
Brief Title: Immune Regulation in Chronic Aspergillus Infection After COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2023-01-002BC
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood test will be obtained within first 3 months, 3-6 months, and 12 months after anticipates agree to enrolled into the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aspergillosis: Patients with aspergillosis
  Interventions: Other: This is a blood test without regarding to intervention nor diagnostic tests
- COVID: Patients with history of COVID infection and without aspergillosis
  Interventions: Other: This is a blood test without regarding to intervention nor diagnostic tests
- Control: Patients without history of COVID infection and without aspergillosis
  Interventions: Other: This is a blood test without regarding to intervention nor diagnostic tests

INTERVENTIONS:
Other: This is a blood test without regarding to intervention nor diagnostic tests — This is a blood test without regarding to intervention nor diagnostic tests

SUMMARY:
This study aims to collect clinical cases and follow-up data from patients with chronic pulmonary aspergillosis, post-COVID-19 aspergillosis, and post-COVID-19 patients without aspergillosis. Using in vitro assays, we will measure the phagocytic function of neutrophils when stimulated by fungal hyphae, their ability to produce neutrophil extracellular traps (NETs), the expression of cell surface molecules at the time of enrollment, changes in cell surface molecule expression after stimulation with fungal hyphae, and the quantification of autoantibodies in the blood. This research will focus on the short-term (within 3 months), medium-term (6-12 months), and long-term (more than 12 months) changes in cell surface molecules and functions following infection.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases include patients diagnosed with pulmonary aspergillosis, acute or subacute Aspergillus infections, and aspergillosis in other anatomical sites (such as sinuses, middle ear, liver). Additionally, this study will enroll patients with chronic obstructive pulmonary disease (COPD), asthma, or those undergoing treatment for pulmonary tuberculosis who continue to exhibit worsening pulmonary radiological findings without a clear etiology, necessitating hospitalization or outpatient care for unexplained community-acquired pneumonia. Patients with bronchiectasis, emphysema, pulmonary fibrosis, or other chronic pulmonary conditions who are under continuous follow-up and treatment at our institution will also be included if clinically diagnosed with aspergillosis.

The control group will consist of patients who, based on clinical evidence, have no history of prior exposure to Aspergillus or aspergillosis infection after contracting COVID-19.

Exclusion Criteria:

* Individuals aged below 20, pregnant women, patients with advanced-stage (stage II and above) lung cancer, individuals diagnosed with malignancies, patients with mental health disorders requiring consent from a legal guardian for participation, and those in critical end-stage conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients with and without COVID infection, and with aspergillus coinfection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months intervel
  The study will observed for at least one year for overall survival

SECONDARY OUTCOMES:
Oppertunistic infection | yearly
  Infection not by aspergillus or COVID

CONTACTS AND LOCATIONS:
Overall Officials: SF Huang, Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Shiang Fen Huang, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No